CLINICAL TRIAL: NCT04693481
Title: Effects of Nature Exposure Intervention on Self-Regulation and Decision-making in Mentally Fatigued University Soccer Players
Brief Title: Effects of Nature Exposure Intervention on Soccer Performance Among Mentally Fatigued University Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Sun He, Principal investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JKEUPM-2020-327
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Mental Fatigue
Keywords: decision-making skills; self-regulation; mental fatigue; soccer performance
MeSH Terms: conditions — Mental Fatigue; Self-Control

STUDY DESIGN:
Intervention Model Description: Randomly assign subjects into the experimental groups and the control group
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- experimental group: 5 seconds for each photo (Experimental): receive the intervention, which is viewing each nature photo for 5 seconds
  Interventions: Other: nature exposure
- experimental group: 15 seconds for each photo (Experimental): receive the intervention, which is viewing each nature photo for 15 seconds
  Interventions: Other: nature exposure
- experimental group: 30 seconds for each photo (Experimental): receive the intervention, which is viewing each nature photo for 30 seconds
  Interventions: Other: nature exposure
- control group (No Intervention): not receive the intervention, which is viewing each nature photo for 0 seconds.

INTERVENTIONS:
Other: nature exposure — Nature exposure has different ways, such as walk in the real nature environment; viewing nature photos. Two main reasons make this study will not use the real nature environment: (1) the limitation of time before or amid the soccer competition; (2) the pandemic situation does not allow people go outside as frequently as before. Therefore, the current study will select some nature photos, which are restorative environments and can restore directed attention to counteract mental fatigue.
  Arms: experimental group: 15 seconds for each photo; experimental group: 30 seconds for each photo; experimental group: 5 seconds for each photo

SUMMARY:
The current study is going to investigate the nature exposure intervention on the ability of self-regulation and decision-making skills among mentally fatigued soccer players. The subjects will be instructed to view some nature photos, which can facilitate the recovering process for directed attention and the ability of self-regulation. Thus, to see the improvement in decision-making skills.

DETAILED DESCRIPTION:
The intervention of this study is nature exposure, specifically, instruct subjects to view and immerse in some nature photos due to the humanity of biophilia.

The condition of mental fatigue will be induced by the Stroop task.

Before the intervention or process of viewing photos, the baseline will be recorded to compare the post-test value of self-regulation and the score of decision-making skills.

Moreover, the different durations of viewing photos will be implemented to identify the optimal selection.

ELIGIBILITY:
Inclusion Criteria:

* The selection of the participants will be every position without the goalkeeper. The age of them will be at 18-24 years. Only male players will be selected. Players should have at least played from the senior school and have 3 years' training experience.

Exclusion Criteria:

* The study will exclude color blindness, for the Stroop task will involve color. Self-reports should be free of any known disease or sleep disorder and not currently taking any medication.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) will be the indicator of physiological self-regulation and measured by Polar H10 HRV belt | 2 weeks
  Before and after the intervention, the HRV will be measured to see the differences.
State anxiety will be the indicator of psychological self-regulation and measured by Competitive State Anxiety Inventory-2 | 2 weeks
  Before and after the intervention, the state anxiety will be measured to see the differences. The arrange of scores of Competitive State Anxiety Inventory-2 is 9-36. The higher scores mean higher cognitive and physical anxiety, as well as state confidence.
The soccer decision-making skills will be measured by TacticUP soccer performance online system | 2 weeks
  Before and after the intervention, the decision-making skills will be measured to see the differences. The arrange of score in TacticUp is 0-100. The higher score, the better decision-making skill.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun He, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided